CLINICAL TRIAL: NCT05173051
Title: Medication Intake of Solid Dosage Forms: A Risk Factor for Patients With Stroke-induced Dysphagia?
Acronym: MedISID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Michaela Trapl-Grundschober, Principal Investigator, Karl Landsteiner University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11TS003721
Record Dates: First submitted 2021-12-13; First posted 2021-12-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Infarction; Stroke, Acute; Stroke; Dysphagia
Keywords: Stroke, Acute; Cerebral Infarction; acute first insult; medication intake in dysphagia; Dysphagia; pill dysphagia
MeSH Terms: conditions — Cerebral Infarction; Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ability of Swallowing solid placebos vs. a crushed placebo (Experimental): During routine FEES examination, patients are sequentially being given 3 different solid placebos pills and one crushed placebo mixed with semisolid texture.
  Interventions: Other: Solid Medication intake vs. crushed medication intake

INTERVENTIONS:
Other: Solid Medication intake vs. crushed medication intake — The swallowing ability for solid and crushed medications in stroke patients is evaluated.
  Other Names: Medication Intake of Solid Dosage Forms

SUMMARY:
In a prospective, quantitative explorative study, the risk of aspiration and penetration when swallowing solid pills (placebo) compared to a crushed placebo pill will be evaluated during a routine Fiberoptic Endoscopic Evaluation of Swallowing (FEES). The study design is thus a quasi-experimental study design with repeated measurements in the sense of a pre-posttest. Each patient undergoes a baseline examination (routine procedure) followed by the intervention (administration of three different solid pills and a crushed pill).

DETAILED DESCRIPTION:
In the research landscape, the topic of medication intake in patients with dysphagia has generally received very little attention, which is why hardly any recommendations can be found in the current guidelines. In the national guidelines of the National Institute for Health and Care Excellence (NICE), the following paragraph was added in 2019: "People with acute stroke who are unable to take adequate nutrition, fluids and medication orally should have their oral medication reviewed to amend either the formulation or the route of administration". In the studies by Kelly and colleagues, dysphagia patients were up to three times more likely to receive an erroneous medication administration than patients without dysphagia. It is therefore currently completely unclear how solid medications can be administered safely in patients with acute dysphagia. There is a complete lack of scientific research in this area which means that the way solid medications are administered to patients with dysphagia is based solely on medical and/or nursing experience.

In everyday clinical practice, solid medications are often delivered in a crushed form to make them easier for patients to swallow. This practice is not evidence-based and has no scientific foundation. There is not a single study known to the author that has systematically investigated the swallowability of crushed medications using an instrumental procedure. Thus, there is an urgent need for research to investigate whether crushed pills can be swallowed better than solid medications by using semisolid textures. This research focuses mainly on the stroke population.

Research questions:

Based on the current state of research and the research gap presented, an overarching research question emerges: "Do patients with acute stroke and recent dysphagia also have a swallowing dysfunction for solid medications? Two subprojects are planned to answer the overall research question: A questionnaire analysis and a clinical experimental study.

The questionnaire analysis serves as a first orientation on how the topic is handled on the stroke units. One question in the questionnaire is aimed at finding out which bolus is most frequently used for the administration of medication. The clinical trial is then conducted with this result.

In a clinical quasi-experimental study, the swallowing ability of placebo medication in patients with dysphagia will be assessed using Fiberoptic Endoscopic Evaluation of Swallowing (FEES).

Primary research question "Questionnaire study" "How is medication administration on stroke units, based on dysphagia screening currently performed?" Primary research questions "Clinical study" Is there a different aspiration-penetration risk when swallowing solid medication and when swallowing crushed medication?

Methods:

In a prospective, quantitative explorative study, the risk of aspiration and penetration when swallowing solid pills (placebo) compared to a crushed placebo pill will be evaluated during a routine Fiberoptic Endoscopic Swallowing Examination (FEES). The study design is thus a quasi-experimental study design with repeated measurements in the sense of a pre-posttest. Each patient undergoes a baseline examination (routine procedure) followed by the intervention (administration of three different solid pills and a crushed pill). Randomisation is not foreseen in a quasi-experimental study or in an evaluation study.

Inclusion/exclusion criteria In this part of the study, 60 patients between 50 and 90 years of age who are admitted to the stroke unit of the neurology department at the University Hospital Tulln with an acute first insult, who have a GUSS result of less than 20 points, and who give written consent to participate in the study, are consecutively included. In addition, there must be a need for endoscopy, based on the screening result and the clinical swallowing examination.

All patients with additional neurodegenerative diseases, with re-insult, all patients in the time window of 2 hours after extubation, tracheotomy, COPD, patients with pre-existing dysphagia and with pre-existing swallowing problems with tablet swallowing are excluded. All patients who are not eligible for swallow endoscopy are also excluded.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 50 and 90 years of age who are admitted to the stroke unit of the neurology department at the University Hospital of Tulln with an acute first stroke, who have a Gugging Swallowing Screen (GUSS) result of less than 20 points, and who give written consent to participate in the study, are consecutively included. In addition, there must be a need for endoscopy (FEES), based on the screening result and the clinical swallowing examination.

Exclusion Criteria:

* All patients with additional neurodegenerative diseases, with re-stroke, all patients in the time window of 2 hours after extubation, tracheostomy, chronic obstructive pulmonary disease (COPD), patients with pre-existing dysphagia and with pre-existing tablet swallowing problems are excluded. All patients who are not eligible for FEES (Fiberoptic Endoscopic Evaluation of Swallowing) are also excluded. This includes the following diagnoses: Skull base fractures / facial fractures, severe, life-threatening epistaxis in the last 6 weeks, nasal cavity trauma, nasal and paranasal surgery, nasal and paranasal injury in the last 6 weeks, sinus nasal tumours, skull base tumours / surgery, nasopharyngeal stenoses, craniofacial anomalies, Osler's disease (hereditary haemorrhagic telangiectasia), known vasovagal episodes.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale (PAS) ≥ 3 for each solid placebo and for the crushed placebo in comparison. | Immediately after the intervention
  Penetration Aspiration Scale (PAS) is measured during the Swallow endoscopy (FEES). The PAS is a measure of the penetration and aspiration of a bolus.
  Scala ranges from 1-8.
  1. Material does not enter the airway
  2. Material enters the airway, remains above the vocal folds, and is ejected from the airway
  3. Material enters the airway, remains above the vocal folds, and is not ejected from the airway
  4. Material enters the airway, contacts the vocal folds, and is ejected from the airway
  5. Material enters the airway, contacts the vocal folds, and is not ejected from the airway
  6. Material enters the airway, passes below the vocal folds and is ejected into the larynx or out of the airway
  7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort
  8. Material enters the airway, passes below the vocal folds, and no effort is made to eject
Penetration Aspiration Scale (PAS) ≥ 3 for the accompanying bolus | Immediately after the intervention
  Penetration Aspiration Scale (PAS) is measured during the Swallow endoscopy (FEES). The PAS is a measure of the penetration and aspiration of a bolus.
  Scala ranges from 1-8.
  1. Material does not enter the airway
  2. Material enters the airway, remains above the vocal folds, and is ejected from the airway
  3. Material enters the airway, remains above the vocal folds, and is not ejected from the airway
  4. Material enters the airway, contacts the vocal folds, and is ejected from the airway
  5. Material enters the airway, contacts the vocal folds, and is not ejected from the airway
  6. Material enters the airway, passes below the vocal folds and is ejected into the larynx or out of the airway
  7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort
  8. Material enters the airway, passes below the vocal folds, and no effort is made to eject

SECONDARY OUTCOMES:
FEES-based graduation of ability to swallow oral solid medication | Immediately after the intervention
  This is a 4 point severity rating scale modified after Buhmann et al. 2019

CONTACTS AND LOCATIONS:
Overall Officials: Walter Struhal, Prof. Dr, Study Chair — University Clinic Tulln
Locations (1):
- University Clinic Tulln, Tulln, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Khaled M, Matthis C, Binder A, Mudter J, Schattschneider J, Pulkowski U, Strohmaier T, Niehoff T, Zybur R, Eggers J, Valdueza JM, Royl G; for QugSS II Group. Dysphagia in Patients with Acute Ischemic Stroke: Early Dysphagia Screening May Reduce Stroke-Related Pneumonia and Improve Stroke Outcomes. Cerebrovasc Dis. 2016;42(1-2):81-9. doi: 10.1159/000445299. Epub 2016 Apr 13. PMID 27074007
- [Background] Arnold M, Liesirova K, Broeg-Morvay A, Meisterernst J, Schlager M, Mono ML, El-Koussy M, Kagi G, Jung S, Sarikaya H. Dysphagia in Acute Stroke: Incidence, Burden and Impact on Clinical Outcome. PLoS One. 2016 Feb 10;11(2):e0148424. doi: 10.1371/journal.pone.0148424. eCollection 2016. PMID 26863627
- [Background] Baijens LW, Clave P, Cras P, Ekberg O, Forster A, Kolb GF, Leners JC, Masiero S, Mateos-Nozal J, Ortega O, Smithard DG, Speyer R, Walshe M. European Society for Swallowing Disorders - European Union Geriatric Medicine Society white paper: oropharyngeal dysphagia as a geriatric syndrome. Clin Interv Aging. 2016 Oct 7;11:1403-1428. doi: 10.2147/CIA.S107750. eCollection 2016. PMID 27785002
- [Background] Bray BD, Smith CJ, Cloud GC, Enderby P, James M, Paley L, Tyrrell PJ, Wolfe CD, Rudd AG; SSNAP Collaboration. The association between delays in screening for and assessing dysphagia after acute stroke, and the risk of stroke-associated pneumonia. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):25-30. doi: 10.1136/jnnp-2016-313356. Epub 2016 Jun 13. PMID 27298147
- [Background] Buhmann C, Bihler M, Emich K, Hidding U, Potter-Nerger M, Gerloff C, Niessen A, Flugel T, Koseki JC, Nienstedt JC, Pflug C. Pill swallowing in Parkinson's disease: A prospective study based on flexible endoscopic evaluation of swallowing. Parkinsonism Relat Disord. 2019 May;62:51-56. doi: 10.1016/j.parkreldis.2019.02.002. Epub 2019 Feb 4. PMID 30770254
- [Background] Carnaby-Mann G, Crary M. Pill swallowing by adults with dysphagia. Arch Otolaryngol Head Neck Surg. 2005 Nov;131(11):970-5. doi: 10.1001/archotol.131.11.970. PMID 16301368
- [Background] CARRIER, M. 2019. Wissenschaftstheorie zur Einführung, Junius Verlag.
- [Background] Cichero JA. Thickening agents used for dysphagia management: effect on bioavailability of water, medication and feelings of satiety. Nutr J. 2013 May 1;12:54. doi: 10.1186/1475-2891-12-54. PMID 23634758
- [Background] Cichero JA, Lam P, Steele CM, Hanson B, Chen J, Dantas RO, Duivestein J, Kayashita J, Lecko C, Murray J, Pillay M, Riquelme L, Stanschus S. Development of International Terminology and Definitions for Texture-Modified Foods and Thickened Fluids Used in Dysphagia Management: The IDDSI Framework. Dysphagia. 2017 Apr;32(2):293-314. doi: 10.1007/s00455-016-9758-y. Epub 2016 Dec 2. PMID 27913916
- [Background] Marquis J, Schneider MP, Payot V, Cordonier AC, Bugnon O, Hersberger KE, Arnet I. Swallowing difficulties with oral drugs among polypharmacy patients attending community pharmacies. Int J Clin Pharm. 2013 Dec;35(6):1130-6. doi: 10.1007/s11096-013-9836-2. Epub 2013 Aug 21. PMID 23963541
- [Background] DÖRING, N. & BORTZ, J. 2016. Forschungsmethoden und Evaluation. Wiesbaden: Springerverlag.
- [Background] Dziewas R, Auf dem Brinke M, Birkmann U, Brauer G, Busch K, Cerra F, Damm-Lunau R, Dunkel J, Fellgiebel A, Garms E, Glahn J, Hagen S, Held S, Helfer C, Hiller M, Horn-Schenk C, Kley C, Lange N, Lapa S, Ledl C, Lindner-Pfleghar B, Mertl-Rotzer M, Muller M, Neugebauer H, Ozsucu D, Ohms M, Perniss M, Pfeilschifter W, Plass T, Roth C, Roukens R, Schmidt-Wilcke T, Schumann B, Schwarze J, Schweikert K, Stege H, Theuerkauf D, Thomas RS, Vahle U, Voigt N, Weber H, Werner CJ, Wirth R, Wittich I, Woldag H, Warnecke T. Safety and clinical impact of FEES - results of the FEES-registry. Neurol Res Pract. 2019 Apr 26;1:16. doi: 10.1186/s42466-019-0021-5. eCollection 2019. PMID 33324882
- [Background] DZIEWAS, R. & PFLUG, C. 2020. Neurogene Dysphagie, S1-Leitlinie, 2020 [Online]. Deutsche Gesellschaft für Neurologie (Hrsg.) Available: www.dgn.org/leitlinien [Accessed 2020].
- [Background] Fields J, Go JT, Schulze KS. Pill Properties that Cause Dysphagia and Treatment Failure. Curr Ther Res Clin Exp. 2015 Aug 20;77:79-82. doi: 10.1016/j.curtheres.2015.08.002. eCollection 2015 Dec. PMID 26543509
- [Background] Forough AS, Lau ET, Steadman KJ, Cichero JA, Kyle GJ, Serrano Santos JM, Nissen LM. A spoonful of sugar helps the medicine go down? A review of strategies for making pills easier to swallow. Patient Prefer Adherence. 2018 Jul 26;12:1337-1346. doi: 10.2147/PPA.S164406. eCollection 2018. PMID 30100710
- [Background] Fujishima I, Fujiu-Kurachi M, Arai H, Hyodo M, Kagaya H, Maeda K, Mori T, Nishioka S, Oshima F, Ogawa S, Ueda K, Umezaki T, Wakabayashi H, Yamawaki M, Yoshimura Y. Sarcopenia and dysphagia: Position paper by four professional organizations. Geriatr Gerontol Int. 2019 Feb;19(2):91-97. doi: 10.1111/ggi.13591. Epub 2019 Jan 9. PMID 30628181
- [Background] FUSCO, S., CARIATI, D., SCHEPISI, R., GANZETTI, R., SESTILI, M., DAVID, S., FERRARA, L., GATTO, M. L., VENA, S., CORSONELLO, A. & CORICA, F. 2016. Management of oral drug therapy in elderly patients with dysphagia. Journal of Gerontology and Geriatrics, 64, 9.
- [Background] Gerschke M, Schottker-Koniger T, Forster A, Netzebandt JF, Beushausen UM. Validation of the German Version of the Yale Pharyngeal Residue Severity Rating Scale. Dysphagia. 2019 Jun;34(3):308-314. doi: 10.1007/s00455-018-9935-2. Epub 2018 Aug 16. PMID 30116884
- [Background] GODMAN, H. 2014. Two tricks to make it easier to swallow pills - Harvard Health Blog [Online]. Available: https://www.health.harvard.edu/blog/two-tricks-make-easier-swallow-pills-201411137515 [Accessed].
- [Background] GOLDMAN, A. I. 1997. Science, publicity, and consciousness. Philosophy of Science, 64, 525-545.
- [Background] Griffith R. District nurses' role in managing medication dysphagia. Br J Community Nurs. 2016 Aug 2;21(8):411-5. doi: 10.12968/bjcn.2016.21.8.411. PMID 27479856
- [Background] HEMPEL, C. G. 1958. The theoretician's dilemma: A study in the logic of theory construction.
- [Background] HEMPEL, C. G. 1966. Scientific explanation, Voice of America.
- [Background] Hey C, Pluschinski P, Zaretsky Y, Almahameed A, Hirth D, Vaerst B, Wagenblast J, Stover T. [Penetration-Aspiration Scale according to Rosenbek. Validation of the German version for endoscopic dysphagia diagnostics]. HNO. 2014 Apr;62(4):276-81. doi: 10.1007/s00106-013-2815-z. German. PMID 24633378
- [Background] JACKSON, J. & NAUNTON, M. 2017. Optimising medicine administration in patients with swallowing difficulties. Australian Pharmacist, Education Extra
- [Background] Kelly J, D'Cruz G, Wright D. A qualitative study of the problems surrounding medicine administration to patients with dysphagia. Dysphagia. 2009 Mar;24(1):49-56. doi: 10.1007/s00455-008-9170-3. Epub 2008 Aug 8. PMID 18688675
- [Background] Kelly J, Wright D. Administering medication to adult patients with dysphagia. Nurs Stand. 2009 Mar 25-31;23(29):62-8. doi: 10.7748/ns2009.03.23.29.62.c6928. PMID 19385403
- [Background] Kelly J, Wright D. Administering medication to adult patients with dysphagia: part 2. Nurs Stand. 2010 Mar 3-9;24(26):61-8. PMID 20373615
- [Background] Kelly J, Wright D, Wood J. Medicine administration errors in patients with dysphagia in secondary care: a multi-centre observational study. J Adv Nurs. 2011 Dec;67(12):2615-27. doi: 10.1111/j.1365-2648.2011.05700.x. Epub 2011 May 25. PMID 21615463
- [Background] Kelly J, Wright D, Wood J. Medication errors in patients with dysphagia. Nurs Times. 2012 May 22-28;108(21):12-4. PMID 22774363
- [Background] KEUTH, H. 2013. Karl Popper: Logik der Forschung, Akademie Verlag.
- [Background] Kind A, Anderson P, Hind J, Robbins J, Smith M. Omission of dysphagia therapies in hospital discharge communications. Dysphagia. 2011 Mar;26(1):49-61. doi: 10.1007/s00455-009-9266-4. Epub 2010 Jan 23. PMID 20098999
- [Background] Klotz AL, Zajac M, Ehret J, Hassel AJ, Rammelsberg P, Zenthofer A. Development of a German version of the Oral Health Assessment Tool. Aging Clin Exp Res. 2020 Jan;32(1):165-172. doi: 10.1007/s40520-019-01158-x. Epub 2019 Mar 7. PMID 30847843
- [Background] Lau ETL, Steadman KJ, Cichero JAY, Nissen LM. Dosage form modification and oral drug delivery in older people. Adv Drug Deliv Rev. 2018 Oct;135:75-84. doi: 10.1016/j.addr.2018.04.012. Epub 2018 Apr 13. PMID 29660383
- [Background] Liu F, Ghaffur A, Bains J, Hamdy S. Acceptability of oral solid medicines in older adults with and without dysphagia: A nested pilot validation questionnaire based observational study. Int J Pharm. 2016 Oct 30;512(2):374-381. doi: 10.1016/j.ijpharm.2016.03.007. Epub 2016 Mar 9. PMID 26970368
- [Background] Manrique YJ, Lee DJ, Islam F, Nissen LM, Cichero JA, Stokes JR, Steadman KJ. Crushed tablets: does the administration of food vehicles and thickened fluids to aid medication swallowing alter drug release? J Pharm Pharm Sci. 2014;17(2):207-19. doi: 10.18433/j39w3v. PMID 24934549
- [Background] MARLIANI, B. 2014. Medikamentenassoziierte Schluckstörungen. 4, 18-21.
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Masilamoney M, Dowse R. Knowledge and practice of healthcare professionals relating to oral medicine use in swallowing-impaired patients: a scoping review. Int J Pharm Pract. 2018 Jun;26(3):199-209. doi: 10.1111/ijpp.12447. Epub 2018 Apr 16. PMID 29659107
- [Background] Mc Gillicuddy A, Crean AM, Kelly M, Sahm L. Oral medicine modification for older adults: a qualitative study of nurses. BMJ Open. 2017 Dec 14;7(12):e018151. doi: 10.1136/bmjopen-2017-018151. PMID 29247094
- [Background] MOSES, G. 2020. Don´t take your medicine with fruit juice. MIMS Matters.
- [Background] Neubauer PD, Rademaker AW, Leder SB. The Yale Pharyngeal Residue Severity Rating Scale: An Anatomically Defined and Image-Based Tool. Dysphagia. 2015 Oct;30(5):521-8. doi: 10.1007/s00455-015-9631-4. Epub 2015 Jun 7. PMID 26050238
- [Background] O'HARA, M. 2015. Considerations for medication in dysphagic stroke patients. BJNN/ Stroke Association Supplement.
- [Background] Onder G, Liperoti R, Fialova D, Topinkova E, Tosato M, Danese P, Gallo PF, Carpenter I, Finne-Soveri H, Gindin J, Bernabei R, Landi F; SHELTER Project. Polypharmacy in nursing home in Europe: results from the SHELTER study. J Gerontol A Biol Sci Med Sci. 2012 Jun;67(6):698-704. doi: 10.1093/gerona/glr233. Epub 2012 Jan 4. PMID 22219520
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Prendergast V, Hinkle JL. Oral Care Assessment Tools and Interventions After Stroke. Stroke. 2018 Apr;49(4):e153-e156. doi: 10.1161/STROKEAHA.117.017045. Epub 2018 Mar 13. No abstract available. PMID 29535269
- [Background] PROSIEGEL, M. & WEBER, S. 2013. Dysphagie : Diagnostik und Therapie ; ein Wegweiser für kompetentes Handeln ; [+Online-Material].
- [Background] Qawasmeh MA, Aldabbour B, Momani A, Obiedat D, Alhayek K, Kofahi R, Yassin A, El-Salem K. Epidemiology, Risk Factors, and Predictors of Disability in a Cohort of Jordanian Patients with the First Ischemic Stroke. Stroke Res Treat. 2020 Jun 4;2020:1920583. doi: 10.1155/2020/1920583. eCollection 2020. PMID 32566121
- [Background] RENTELN-KRUSE, W., FRILLING, B., NEUMANN, L. & KUHLMEY, A. 2014. Arzneimittel im Alter.
- [Background] Rofes L, Muriana D, Palomeras E, Vilardell N, Palomera E, Alvarez-Berdugo D, Casado V, Clave P. Prevalence, risk factors and complications of oropharyngeal dysphagia in stroke patients: A cohort study. Neurogastroenterol Motil. 2018 Mar 23:e13338. doi: 10.1111/nmo.13338. Online ahead of print. PMID 29573064
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] SCHAAR, K. 2016. Was hat die Wissenschaft beim Datenschutz künftig zu beachten? Allgemeine und spezifische Änderungen beim Datenschutz im Wissenschaftsbereich durch die neue Europäische Datenschutzgrundverordnung. RatSWD Working Paper.
- [Background] Schiele JT, Penner H, Schneider H, Quinzler R, Reich G, Wezler N, Micol W, Oster P, Haefeli WE. Swallowing Tablets and Capsules Increases the Risk of Penetration and Aspiration in Patients with Stroke-Induced Dysphagia. Dysphagia. 2015 Oct;30(5):571-82. doi: 10.1007/s00455-015-9639-9. Epub 2015 Jul 24. PMID 26205435
- [Background] Schiele JT, Schneider H, Quinzler R, Reich G, Haefeli WE. Two techniques to make swallowing pills easier. Ann Fam Med. 2014 Nov-Dec;12(6):550-2. doi: 10.1370/afm.1693. PMID 25384817
- [Background] SCHNELL, M. W., DUNGER, C. & BARTHOLOMEYCZIK, S. 2018. Forschungsethik: Informieren - reflektieren - anwenden, Hogrefe.
- [Background] Schwemmle C, Jungheim M, Miller S, Kuhn D, Ptok M. [Medication-induced dysphagia : A review]. HNO. 2015 Jul;63(7):504-10. doi: 10.1007/s00106-015-0015-8. German. PMID 26148562
- [Background] Tahaineh L, Wazaify M. Difficulties in swallowing oral medications in Jordan. Int J Clin Pharm. 2017 Apr;39(2):373-379. doi: 10.1007/s11096-017-0449-z. Epub 2017 Mar 9. PMID 28281225
- [Background] Takizawa C, Gemmell E, Kenworthy J, Speyer R. A Systematic Review of the Prevalence of Oropharyngeal Dysphagia in Stroke, Parkinson's Disease, Alzheimer's Disease, Head Injury, and Pneumonia. Dysphagia. 2016 Jun;31(3):434-41. doi: 10.1007/s00455-016-9695-9. Epub 2016 Mar 12. PMID 26970760
- [Background] Trapl M, Enderle P, Nowotny M, Teuschl Y, Matz K, Dachenhausen A, Brainin M. Dysphagia bedside screening for acute-stroke patients: the Gugging Swallowing Screen. Stroke. 2007 Nov;38(11):2948-52. doi: 10.1161/STROKEAHA.107.483933. Epub 2007 Sep 20. PMID 17885261
- [Background] TRAPL-GRUNDSCHOBER, M. 2017. Bevölkerungsgesundheitliche Bedeutung der Identifikation von Risikofaktoren für die Entwicklung von Schluckstörungen im Rahmen des physiologischen Alterungsprozesses. Eine Stichprobenanalyse. PhDr. Doktorarbeit, Universität für Gesundheit und Sozialarbeit St. Alžbety Bratislava.
- [Background] Wakabayashi H. Presbyphagia and Sarcopenic Dysphagia: Association between Aging, Sarcopenia, and Deglutition Disorders. J Frailty Aging. 2014;3(2):97-103. doi: 10.14283/jfa.2014.8. PMID 27049901
- [Background] Wakabayashi H, Takahashi R, Murakami T. The Prevalence and Prognosis of Sarcopenic Dysphagia in Patients Who Require Dysphagia Rehabilitation. J Nutr Health Aging. 2019;23(1):84-88. doi: 10.1007/s12603-018-1117-2. PMID 30569074
- [Background] Warnecke T, Im S, Kaiser C, Hamacher C, Oelenberg S, Dziewas R. Aspiration and dysphagia screening in acute stroke - the Gugging Swallowing Screen revisited. Eur J Neurol. 2017 Apr;24(4):594-601. doi: 10.1111/ene.13251. Epub 2017 Feb 3. PMID 28322006
- [Background] WHO 2017. WHO | Stroke: a global response is needed. WHO.
- [Background] WHO 2018. WHO | Global Health Estimates. WHO.
- [Background] Yin OQ, Rudoltz M, Galetic I, Filian J, Krishna A, Zhou W, Custodio J, Golor G, Schran H. Effects of yogurt and applesauce on the oral bioavailability of nilotinib in healthy volunteers. J Clin Pharmacol. 2011 Nov;51(11):1580-6. doi: 10.1177/0091270010384116. Epub 2011 Jun 28. PMID 21712497
- [Background] Zhao WT, Yang M, Wu HM, Yang L, Zhang XM, Huang Y. Systematic Review and Meta-Analysis of the Association between Sarcopenia and Dysphagia. J Nutr Health Aging. 2018;22(8):1003-1009. doi: 10.1007/s12603-018-1055-z. PMID 30272106
- [Derived] Trapl-Grundschober M, Struhal W, Teuschl Y, Schulz S, Sollereder S, Osterbrink J. Medication Administration in Poststroke Dysphagia: Evaluating Swallowing Safety of Solid Dosage Forms. Stroke. 2025 Sep;56(9):2494-2502. doi: 10.1161/STROKEAHA.125.051237. Epub 2025 Jul 16. PMID 40665903
- [Derived] Trapl-Grundschober M, Schneider L, Schulz S, Sollereder S, Teuschl Y, Struhal W, Osterbrink J. Solid Medication Intake in Hospitalised Patients With Dysphagia: A Challenge for Speech and Language Pathologists? Int J Lang Commun Disord. 2025 Jul-Aug;60(4):e70073. doi: 10.1111/1460-6984.70073. PMID 40605450
- [Derived] Trapl-Grundschober M, Schulz S, Sollereder S, Schneider L, Teuschl Y, Osterbrink J. Oral intake of solid medications in patients with post-stroke dysphagia. A challenge for nurses? J Clin Nurs. 2025 Mar;34(3):872-882. doi: 10.1111/jocn.17081. Epub 2024 Feb 26. PMID 38407372
- See also: NICEGUIDLINE (NG128). 2019. Stroke and transient ischaemic attack in over 16s: diagnosis and initial management [Online]. Available: — https://www.nice.org.uk/guidance/ng128/chapter/Recommendations#avoiding-aspiration-pneumonia
- See also: Tips for Swallowing Pills [Online] OSMAN, J. 2017. Available: [Accessed]. — https://caregiver.com/api/content/2c5fb0a2-3580-11e7-8125-0aea2a882f79/
- See also: THE NATIONAL LIBRARY OF MEDICINE. 2020. ClinicalTrials.gov [Online]. Available:[Accessed]. — https://www.clinicaltrials.gov/ct2/home
- See also: Research Randomizer [Online] URBANIAK, G. C. & PLOUS, S. 2020. Available: — https://www.randomizer.org